CLINICAL TRIAL: NCT07345312
Title: The Use of the BodySleep Algorithm (ResMed) for the Diagnosis of Obstructive Sleep Apnea Syndrome in Children
Brief Title: BodySleep Algorithm for OSA Diagnosis in Children
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PI030
Record Dates: First submitted 2023-03-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea of Child
MeSH Terms: interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Polysomnography — PSG performed prospectively in routine care in children suspected of OSA

SUMMARY:
Diagnosing obstructive sleep apnea-hypopnea syndrome in children (OSA) requires the performance of polysomnography (PSG) in the hospital which is sometimes challenging to perform in children, and time-consuming for installation and analysis. Simplified recording and analysis methods are preferable in children but require validation in this population.

The BodySleep automatic algorithm of the polysomnograph used in our lab (A1-Nox, ResMed) associated only with respiratory signals could be used to identify respiratory events. Thus the child would have fewer sensors installed on him.

DETAILED DESCRIPTION:
The diagnosis of obstructive sleep apnea-hypopnea syndrome in children (OSA) requires the performance of polysomnography (PSG) in the hospital with video surveillance and monitoring by a nurse to put the sensors back on the child if necessary. During the night. The PSG gives the index of obstructive apnea-hypopnea (IAHO) necessary for the diagnosis of OSAS and to determine its severity. But the PSG is a rather cumbersome examination, sometimes challenging to perform in children, with several sensors and electrodes to install (electroencephalogram (EEG), electromyogram (EMG), electrooculogram (EOG), necessary to determine the periods of wakefulness -sleep and intra-sleep micro-arousals, nasal cannula, thoracoabdominal straps, pulse oximetry, actimetry to score respiratory events), time-consuming for installation and analysis. Simplified recording and analysis methods are preferable in children but require validation in this population.

The BodySleep automatic algorithm of the polysomnograph used in our service (A1-Nox, ResMed) combines actigraphy data (body position during sleep) and induction plethysmography signal resulting from the thoracoabdominal belts to identify sleep-wake stages could be used instead of EEG, EOG and EMG electrodes. The BodySleep algorithm associated only with respiratory signals (nasal cannula, thoracoabdominal straps, pulse oximetry, actimetry) could be used to identify respiratory events. Thus the child would have fewer sensors installed on him.

The hypothesis of this study is that the BodySleep algorithm associated with respiratory signals can identify OSA in children.

ELIGIBILITY:
Inclusion Criteria:

* Children suspected of OSA who are addressed for a PSG by the ear nose throat physician, pediatric pulmonologist, neurologist, psychiatrist, sleep specialist, genetics, and nutritionist physician.
* Age between 2 and 18 years

Exclusion Criteria:

* Age under 2 years and over 18 years

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A retrospective study including children aged 2 to 18 years addressed for a PSG.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Obstructive apnea-hypopnea index by BodySleep in comparison with OAHI by PSG | One night
  To determine if the obstructive apnea-hypopnea index (OAHI) obtained by the BodySleep algorithm is underestimated in comparison with the OAHI obtained by the PSG

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dietz-Terjung S, Martin AR, Finnsson E, Agustsson JS, Helgason S, Helgadottir H, Welsner M, Taube C, Weinreich G, Schobel C. Proof of principle study: diagnostic accuracy of a novel algorithm for the estimation of sleep stages and disease severity in patients with sleep-disordered breathing based on actigraphy and respiratory inductance plethysmography. Sleep Breath. 2021 Dec;25(4):1945-1952. doi: 10.1007/s11325-021-02316-0. Epub 2021 Feb 16. PMID 33594617